CLINICAL TRIAL: NCT03503526
Title: Trauma-focused Group Music and Imagery With Women Suffering From PTSD/Complex PTSD
Brief Title: Trauma-focused Group Music and Imagery With Traumatized Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Collaborators: Kris- och Traumacentrum Sverige AB (Unknown); Council of the Danish Victims Fund (Unknown)
Responsible Party: Principal Investigator, Gabriella Rudstam, Principal Investigator, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015/895-31; 15-910-00019 (Other Grant/Funding Number: Council of the Danish Victims Fund)
Record Dates: First submitted 2018-02-19; First posted 2018-04-20 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: A randomized wait list control study with a mixed methods design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music therapy treatment (Experimental): An intervention consisting of 12 weekly sessions of trauma-focused treatment in form of group music and imagery therapy.
  Receptive music therapy.
  Interventions: Behavioral: Receptive music therapy
- Wait List Control (No Intervention): No treatment for approximately 12 weeks.

INTERVENTIONS:
Behavioral: Receptive music therapy — 12 weekly trauma-focused Group therapy sessions of a length of 2.5 hours. The core element is receptive music psychotherapy with music listening, art making, and other art based methods.
  Other Names: Group Music and Imagery and Expressive Arts therapy
  Arms: Music therapy treatment

SUMMARY:
This study is a mixed methods randomized controlled trial (Wait List Control), that investigates the effects of Group Music and Imagery (GrpMI) therapy in the treatment of women suffering from Post Traumatic Stress Disorder (PTSD) or Complex PTSD.

The aim is to detect if the intervention has an effect on PTSD symptoms, dissociation, quality of life, and the capability of regulating the autonomic nervous system (ANS).

DETAILED DESCRIPTION:
Participants are adult women suffering from PTSD or Complex PTSD (n=56) that are randomized to three months of weekly (12) sessions of trauma modified GrpMI therapy or no treatment for an equal amount of time (wait list control).

Primary outcome is pre, post and 3 months follow-up measures of PTSD checklist 5 (PCL-5).

Secondary outcome is pre, post and 3 months follow-up measures of dissociative experience scale (DES), positive state of mind scale (PSOM-S), Hopkins symptoms checklist (HSCL-25), somatoform dissociation questionnaire (SDQ-5), and reactivity and recovery of different physiological measures related to arousal regulation ability in a script driven imagery setting.

ELIGIBILITY:
Inclusion Criteria:

* be suffering from PTSD/CPTSD,
* be sufficiently stabilised to tolerate being exposed to trauma treatment and listen to other subjects' stories,
* be able to speak good enough swedish to express themselves without an interpreter,
* have an interest in working with their problems using artistic languages,
* have an ability to work with symbolism and inner images.

Exclusion Criteria:

* difficulties in understanding or making themselves understood in swedish,
* severe personality disorder or neuropsychiatric disorder,
* ongoing alcohol or drug abuse,
* psychotic disorder,
* suicidality,
* serious ongoing medical condition,
* serious psychosocial problems.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male subjects meeting the inclusion criteria are not readily available at the clinic where the study is conducted.
Enrollment: 45 (Actual)
Dates: Start 2015-08-13 (Actual); Primary Completion 2018-08-22 (Actual); Study Completion 2018-08-22 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Posttraumatic Stress Disorder Checklist (version 5) (PCL-5) total score at 3 months (post intervention) and at 6 months (follow- up). | Baseline, 3 months (post intervention) and 6 months (follow- up).
  PCL-5 is a 20-item self-assessment scale, measuring symptoms related to posttraumatic stress disorder (PTSD). The total score range are from 0-80. Higher scores indicate more severe PTSD symptoms.

SECONDARY OUTCOMES:
Change from baseline in Dissociative experience scale (DES) mean score at 3 months (post intervention) and at 6 months (follow- up). | Baseline, 3 months (post intervention) and 6 months (follow- up).
  DES is a 28-item self-assessment scale that measures psychoform dissociation. Each item ranges from 0 % to 100 % and the mean score is used as an index for the severity of the dissociative symptoms. A higher mean score indicates more dissociative symptoms.
Change from baseline in Hopkins symptom checklist (HSCL-25) mean scores at 3 months (post intervention) and at 6 months (follow- up). | Baseline, 3 months (post intervention) and 6 months (follow- up).
  HSCL-25 is a 25-item self-assessment scale with two subscales. The first subscale measures anxiety and has 10 items. Each item ranges from 1 to 4. The mean score is used as an index of anxiety. A high mean score indicates more anxiety symptoms. The second subscale measures depression and has 15 items. Each item range from 1 to 4. The mean score is used as an index of depression. Higher mean score indicate more depressive symptoms.
Change from baseline in Positive states of mind scale (PSOM-S) total score at 3 months (post intervention) and at 6 months (follow- up). | Baseline, 3 months (post intervention) and 6 months (follow- up).
  PSOM-S is a 5-item self-assessment scale that measures quality of life. The total range are from 5-15. Higher scores indicate a higher quality of life.
Change from baseline in Somatoform Dissociation Questionnaire (SDQ5) total score at 3 months (post intervention) and at 6 months (follow- up). | Baseline, 3 months (post intervention) and 6 months (follow- up).
  SDQ5 is a 5-item self-assessment scale that measures somatoform dissociation. The total range are from 5-15. Higher scores indicates more severe somatoform dissociative symptoms.
Change from baseline in timeline of heart rate during exposure to script-driven trauma imagery at 3 months (post intervention) and 6 months (follow-up). | Baseline, 3 months (post intervention) and 6 months (follow- up).
  Heart rate (bpm) measured with a blood volume pulse sensor.
Change from baseline in timeline of peripheral temperature during exposure to script-driven trauma imagery at 3 months (post intervention) and 6 months (follow-up). | Baseline, 3 months (post intervention) and 6 months (follow- up).
  Temperature measured on the fingertip of the left hand´s middle finger.
Change from baseline in timeline of skin conductance level during exposure to script-driven trauma imagery at 3 months (post intervention) and 6 months (follow-up). | Baseline, 3 months (post intervention) and 6 months (follow- up).
  Measured with electrodes on the proximal phalanges of the left hand´s index and ring finger.
Change from baseline in timeline of muscle tension during exposure to script-driven trauma imagery at 3 months (post intervention) and 6 months (follow-up). | Baseline, 3 months (post intervention) and 6 months (follow- up).
  Measured as root mean square amplitude of the electromyography signal (micro volt) with electrodes placed on the left forearm (over the extensor digitorum muscle).
Change from baseline in timeline of the root mean square of successive differences (RMSSD) in intervals between individual heart beats during exposure to script-driven trauma imagery at 3 months (post intervention) and 6 months (follow-up). | Baseline, 3 months (post intervention) and 6 months (follow- up).
  Derived from the heart rate time series using the beat-to-beat peak blood volume-intervals (measured with a plethysmograph on the right middle finger).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adler NE, Horowitz M, Garcia A, Moyer A. Additional validation of a scale to assess positive states of mind. Psychosom Med. 1998 Jan-Feb;60(1):26-32. doi: 10.1097/00006842-199801000-00006. PMID 9492235
- [Background] First MB. Diagnostic and statistical manual of mental disorders, 5th edition, and clinical utility. J Nerv Ment Dis. 2013 Sep;201(9):727-9. doi: 10.1097/NMD.0b013e3182a2168a. No abstract available. PMID 23995026
- [Background] Bernstein EM, Putnam FW. Development, reliability, and validity of a dissociation scale. J Nerv Ment Dis. 1986 Dec;174(12):727-35. doi: 10.1097/00005053-198612000-00004. PMID 3783140
- [Background] Bovin MJ, Marx BP, Weathers FW, Gallagher MW, Rodriguez P, Schnurr PP, Keane TM. Psychometric properties of the PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders-Fifth Edition (PCL-5) in veterans. Psychol Assess. 2016 Nov;28(11):1379-1391. doi: 10.1037/pas0000254. Epub 2015 Dec 14. PMID 26653052
- [Background] Derogatis LR, Lipman RS, Rickels K, Uhlenhuth EH, Covi L. The Hopkins Symptom Checklist (HSCL): a self-report symptom inventory. Behav Sci. 1974 Jan;19(1):1-15. doi: 10.1002/bs.3830190102. No abstract available. PMID 4808738
- [Background] Horowitz M, Adler N, Kegeles S. A scale for measuring the occurrence of positive states of mind: a preliminary report. Psychosom Med. 1988 Sep-Oct;50(5):477-83. doi: 10.1097/00006842-198809000-00004. PMID 3186891
- [Background] Karatzias T, Shevlin M, Fyvie C, Hyland P, Efthymiadou E, Wilson D, Roberts N, Bisson JI, Brewin CR, Cloitre M. Evidence of distinct profiles of Posttraumatic Stress Disorder (PTSD) and Complex Posttraumatic Stress Disorder (CPTSD) based on the new ICD-11 Trauma Questionnaire (ICD-TQ). J Affect Disord. 2017 Jan 1;207:181-187. doi: 10.1016/j.jad.2016.09.032. Epub 2016 Sep 28. PMID 27723542
- [Background] Koelsch S. A neuroscientific perspective on music therapy. Ann N Y Acad Sci. 2009 Jul;1169:374-84. doi: 10.1111/j.1749-6632.2009.04592.x. PMID 19673812
- [Background] Korlin D, Edman G, Nyback H. Reliability and validity of a Swedish version of the Dissociative Experiences Scale (DES-II). Nord J Psychiatry. 2007;61(2):126-42. doi: 10.1080/08039480701226112. PMID 17454728
- [Background] Nijenhuis ER, Spinhoven P, van Dyck R, van der Hart O, Vanderlinden J. The development of the somatoform dissociation questionnaire (SDQ-5) as a screening instrument for dissociative disorders. Acta Psychiatr Scand. 1997 Nov;96(5):311-8. doi: 10.1111/j.1600-0447.1997.tb09922.x. PMID 9395146
- [Background] Pitman RK, Orr SP, Forgue DF, de Jong JB, Claiborn JM. Psychophysiologic assessment of posttraumatic stress disorder imagery in Vietnam combat veterans. Arch Gen Psychiatry. 1987 Nov;44(11):970-5. doi: 10.1001/archpsyc.1987.01800230050009. PMID 3675137
- [Background] Rudstam G, Elofsson U, Søndergaard HP, Bonde LO, Daniels Beck B. Trauma-focused music and imagery with women suffering from PTSD/complex PTSD: A feasibility study. Approaches: An Interdisciplinary Journal of Music Therapy, Special Issue 9(2): 147-158, 2017.
- [Background] Beck BD, Messell S, Cordtz TO, Sogaard U, Simonsen E, Moe T Feasibility of trauma-focused Guided Imagery and Music with adult refugees diagnosed with PTSD-a pilot study. Nordic Journal of Music Therapy 27(1): 67-86, 2018.
- [Background] Blake R, Bishop S. The Bonny Method of Guided Imagery and Music (GIM) in the Treatment of Post-Traumatic Stress Disorder (PTSD) with Adults in the Psychiatric Setting. Music Therapy Perspectives 12(2): 125-129, 1994.
- [Background] Bruscia K E, Grocke DE. Guided imagery and music: the Bonny method and beyond. Gilsum, NH: Barcelona Pub. 2002.
- [Background] Grocke DE, Moe T (Eds.). Guided imagery & music (GIM) and music imagery methods for individual and group therapy. Philadelphia: Jessica Kingsley Publishers. 2015.
- [Background] Hopper JW, Frewen PA, Sack M, Lanius RA, van der Kolk BA.The Responses to Script-Driven Imagery Scale (RSDI): Assessment of State Posttraumatic Symptoms for Psychobiological and Treatment Research. Journal of Psychopathology and Behavioral Assessment 29(4): 249-268, 2007. https://doi.org/10.1007/s10862-007-9046-0